CLINICAL TRIAL: NCT01465945
Title: A Randomized Clinical Trial of Open Versus Suture Closure in Patients With Rectal Lesions Excised Using Transanal Endoscopic Microsurgery
Brief Title: Study of Unsutured Versus Sutured Closure of Rectal Defects After Rectal Lesion Excisions Using Transanal Endoscopic Microsurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Carl J Brown (Other)
Collaborators: Canadian Society of Colon and Rectal Surgeons (Other)
Responsible Party: Sponsor-Investigator, Dr. Carl J Brown, Head, Division of General Surgery, clinical assistant professor of surgery at University of British Columbia, St. Paul's Hospital, Canada
Organization: St. Paul's Hospital, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TEMPEST
Record Dates: First submitted 2011-10-31; First posted 2011-11-07 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Post-operative Pain; Complications
Keywords: TEM for rectal lesions; Sutured defect; Unsutured defect
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rectal Defect Sutured (Other): The subject will have his/her defect sutured after the rectal tumors have been removed.
  Interventions: Procedure: Defect Sutured
- Rectal Defect Unsutured (Other): The defect will be left open and let naturally close after the rectal tumor has been removed by TEM.
  Interventions: Procedure: Defect Unsutured

INTERVENTIONS:
Procedure: Defect Unsutured — The defect is not sutured after the rectal tumor is removed by TEM.
  Arms: Rectal Defect Unsutured
Procedure: Defect Sutured — Defect is sutured after the rectal tumor has been removed by TEM.
  Arms: Rectal Defect Sutured

SUMMARY:
Transanal Endoscopic Microsurgery (TEM) is a minimally invasive technique used to remove rectal tumours. After the tumour has been removed from the rectum, the surgeon has a choice to close the defect or leave the defect open and naturally close. Currently, both options are accepted as standard care.

Leaving the defect open to close naturally has some possible advantages, including shortened operation time and similar rates of postoperative complications. However, there is some concern that not surgically closing the defect may lead to more postoperative pain and delay in recovery.

The study will be a double blind randomized controlled trial and determine whether patients who have rectal wall defect sutured closed have less post-operative pain compared to patients whose defect is left open.

DETAILED DESCRIPTION:
Summary

Background Transanal Endoscopic Microsurgery (TEM) is an advanced minimally invasive endoluminal technique used to remove rectal tumours. In the open transanal excision era, there is evidence that outcomes in unsutured rectal defects are similar to those in patients whose defect is closed. However, the evidence for this approach is minimal and technical differences in TEM (e.g. rectal insufflation) may mean that leaving defects unsutured is not a safe approach. Further, there is anecdotal evidence that unsutured defects lead to more postoperative pain and delay recovery.

Objective The purpose of this study is to determine if postoperative pain (primary) and early postoperative complications (secondary) are worse in patients undergoing TEM and do not have the defect closed when compare to similar patients who have endoluminal suture closure of the defect.

Methods This is a multicentre, double blind randomized controlled trial of suture closure versus no closure in patients treated by TEM for rectal lesions. The study will include patients 18 years and older with rectal lesions within 12cm of the anal verge treated with TEM. The primary outcome is postoperative pain as measured by validated visual analogue scale (VAS). Secondary outcomes include analgesic use and early (<30 day) complications. Based on anticipated VAS scores, a sample size of 38 patients will be enrolled (power 0.80, α=0.05). Statistical analysis will be performed using student's T test for continuous data and Fischer's exact test for dichotomous variables.

Impact Currently, only 3 centres in Canada have experience with TEM: Vancouver, Winnipeg and Ottawa. This study represents the first trial of a Canadian TEM Collaborative and will determine if there is an advantage to suture closure of the rectal defect in TEM surgery. This is important, as suture technique is challenging and if there are important advantages to this approach, there would be a mandate to perfect suturing technique before employing the TEM approach to rectal tumours. Conversely, if there is an advantage to leaving the defect unsutured, this may reduce operative time and facilitate better use of OR time. Further, it will inform all TEM surgeons of the best approach to the rectal defect and optimize patient care. Finally, this study will serve as a starting point for further trials by the Canadian TEM Collaborative that will expand to include new sites and become a world leader in TEM clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* The patients must be over 18 years old with a rectal lesion < 12cm from the anal verge (as measured by rigid sigmoidoscopy) and less than half the circumference of the rectal lumen. The patient must provide informed consent for TEM and inclusion in the trial.

Exclusion Criteria:

* The surgeon decides to convert to laparotomy or conventional TAE for any reason during tumor excision.
* The surgeon judges that the rectal defect is not appropriate for suturing (e.g. too large) or to be left unsutured (e.g. entry into peritoneal cavity)
* The patient is currently treated for chronic pain prior to surgery, has a known bleeding diathesis (e.g. warfarin treatment, hemophilia, etc) or is immunosuppressed (e.g. Prednisone, HIV,etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 1day after surgery
  As an ancillary measure, all patients will be prescribed 30 tablets of either Tylenol#3 or Tramacet as as their primary postoperative analgesic.

SECONDARY OUTCOMES:
Complications | within 30 days of surgery
  includes bleeding( defined as hemoglobin drop of 20g/L from preoperative and either transfusion, readmission to hospital, or surgical or endoscopic intervention), infection (peritonitis or pelvic pain and either fever >37.9 degC or WBC > 11 X 10^9 c/L), and readmission to hospital for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Brown, MD, MSc, Principal Investigator — Saint Paul's Hospital
Locations (3):
- Canada (3):
  - Saint Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Winnipeg, Manitoba
  - The Ottawa Hospital, Ottawa, Ontario

REFERENCES:
- [Background] McCourt M, Armitage J, Monson JR. Rectal cancer. Surgeon. 2009 Jun;7(3):162-9. doi: 10.1016/s1479-666x(09)80040-1. PMID 19580180
- [Background] Buess G, Hutterer F, Theiss J, Bobel M, Isselhard W, Pichlmaier H. [A system for a transanal endoscopic rectum operation]. Chirurg. 1984 Oct;55(10):677-80. No abstract available. German. PMID 6510078
- [Background] Allaix ME, Arezzo A, Caldart M, Festa F, Morino M. Transanal endoscopic microsurgery for rectal neoplasms: experience of 300 consecutive cases. Dis Colon Rectum. 2009 Nov;52(11):1831-6. doi: 10.1007/DCR.0b013e3181b14d2d. PMID 19966628
- [Background] Ramirez JM, Aguilella V, Arribas D, Martinez M. Transanal full-thickness excision of rectal tumours: should the defect be sutured? a randomized controlled trial. Colorectal Dis. 2002 Jan;4(1):51-55. doi: 10.1046/j.1463-1318.2002.00293.x. PMID 12780656
- [Background] Gallagher EJ, Bijur PE, Latimer C, Silver W. Reliability and validity of a visual analog scale for acute abdominal pain in the ED. Am J Emerg Med. 2002 Jul;20(4):287-90. doi: 10.1053/ajem.2002.33778. PMID 12098173
- [Background] Festen S, van Hoogstraten MJ, van Geloven AA, Gerhards MF. Treatment of grade III and IV haemorrhoidal disease with PPH or THD. A randomized trial on postoperative complications and short-term results. Int J Colorectal Dis. 2009 Dec;24(12):1401-5. doi: 10.1007/s00384-009-0803-2. PMID 19798507
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Kelly AM. The minimum clinically significant difference in visual analogue scale pain score does not differ with severity of pain. Emerg Med J. 2001 May;18(3):205-7. doi: 10.1136/emj.18.3.205. PMID 11354213
- [Background] Burch J, Epstein D, Baba-Akbari A, Weatherly H, Fox D, Golder S, Jayne D, Drummond M, Woolacott N. Stapled haemorrhoidectomy (haemorrhoidopexy) for the treatment of haemorrhoids: a systematic review and economic evaluation. Health Technol Assess. 2008 Apr;12(8):iii-iv, ix-x, 1-193. doi: 10.3310/hta12080. PMID 18373905